CLINICAL TRIAL: NCT04540731
Title: Multicenter Registry of Nonalcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, SEBASTIAN MARCIANO, Assistant Professor of Hepatology, Hospital Italiano de Buenos Aires
Other Study IDs: 5530
Record Dates: First submitted 2020-08-29; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD and diabetes/NASH and fibrosis: Patients with NAFLD and type 2 diabetes (or insulin-resistance) or with any stage of fibrosis in the inclusion visit will be followed over time in a prospective cohort study with scheduled visits. Patients without diabetes/insulin-resistance or any stage of fibrosis will participle in a single visit (inclusion) and will be part of a cross-sectional study.
  Interventions: Other: This is an observational study without intervention
- NAFLD without diabetes/NASH without fibrosis: Patients without diabetes (or insulin-resistance) or any stage of fibrosis will participle in a single visit (inclusion) and will be part of a cross-sectional study
  Interventions: Other: This is an observational study without intervention

INTERVENTIONS:
Other: This is an observational study without intervention — This is an observational study without intervention

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most prevalent liver disease worldwide affecting as much as 25% of the world's population. The spectrum of NAFLD ranges from non-alcoholic fatty liver to non-alcoholic steatohepatitis (NASH), the latter being associated with a progressive course towards fibrosis and a higher risk of developing cirrhosis and hepatocellular carcinoma. Patients with type 2 diabetes are particularly at higher risk of developing fibrosis and advanced liver disease. Since NASH and its consequences will only occur in a minority of patients, it is of paramount importance to identify this population to offer them proper care.

It is well known that there is a lack of awareness about the potential consequences of NAFLD, not only in the general population but also in the medical community. Patients with NAFLD are frequently lost during follow up and, additionally, approach to these patients is sub-optimal and heterogeneous among physicians.

An attractive approach to applying best medical practices to patients with NAFLD is to generate a multicentre registry. Clinical registries comprise a set of systematic collected and stored data focused on a specific condition. The information stored in a registry provides relevant information about a disease and, through a process of error detection, ensures data quality and reliability. A NAFLD registry is an essential tool for providing relevant information such as epidemiological aspects of the disease, outcomes, and treatment effectiveness. As far as we concern, this would be the first registry of NAFLD in our region, a region where the disease behaves in a more aggressive way in comparison with other regions and hemispheres.

By generating this registry, we are confident that we will obtain objective information on the characteristic of patients with NAFLD in our region, not only of the disease characteristics but also of social determinants that might influence disease outcomes. By being a prospective study, it allows an adequate patient follow up.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most prevalent liver disease worldwide affecting as much as 25% of the world's population. The spectrum of NAFLD ranges from non-alcoholic fatty liver to non-alcoholic steatohepatitis (NASH), the latter being associated with a progressive course towards fibrosis and a higher risk of developing cirrhosis and hepatocellular carcinoma. Patients with type 2 diabetes are particularly at higher risk of developing fibrosis and advanced liver disease. Since NASH and its consequences will only occur in a minority of patients, it is of paramount importance to identify this population to offer them proper care.

It is well known that there is a lack of awareness about the potential consequences of NAFLD, not only in the general population but also in the medical community. Patients with NAFLD are frequently lost during follow up and, additionally, approach to these patients is sub-optimal and heterogeneous among physicians.

An attractive approach to applying best medical practices to patients with NAFLD is to generate a multicentre registry. Clinical registries comprise a set of systematic collected and stored data focused on a specific condition. The information stored in a registry provides relevant information about a disease and, through a process of error detection, ensures data quality and reliability. A NAFLD registry is an essential tool for providing relevant information such as epidemiological aspects of the disease, outcomes, and treatment effectiveness. As far as we concern, this would be the first registry of NAFLD in our region, a region where the disease behaves in a more aggressive way in comparison with other regions and hemispheres.

By generating this registry, we are confident that we will obtain objective information on the characteristic of patients with NAFLD in our region, not only of the disease characteristics but also of social determinants that might influence disease outcomes. By being a prospective study, it allows an adequate patient follow up.

With this registry we primarily aim to:

* Describe the characteristics of patients with non-alcoholic fatty liver disease
* Evaluate the disease progression over time (in the sub-group of patients with type 2 diabetes or insulin resistance)
* Identify barriers to achieve best medical practices in non-alcoholic fatty liver disease, such as barriers to adhere to treatment recommendations ,and to access to complementary studies such as elastography or liver biopsy.
* Evaluate patient reported outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 16-year-old)
* NAFLD (defined as proposed by the European Association for the Study of the Liver and the Argentinean Association for the Study of the Liver: "evidence of hepatic steatosis, either by imaging or histology, and lack of secondary causes of liver fat accumulation such as significant alcohol consumption ( >30 g/day for men or > 20 g/day for women), long term use of medications known to cause steatosis, or monogenic hereditary disorders."

Exclusion Criteria:

* Unwillingness to participate in the registry

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with NAFLD.
  In order to properly classify patients with diabetes or insulin resistance, the following criteria will be used:
  -Diabetes: Patients receiving oral anti-diabetic drugs and/or insulin, or who presented a glycated hemoglobin > 6.5 gr/dL or at least 2 fasting glucose levels > 126 mg/dL) Insulin resistance: according to predefined criteria of waist circumference for males and females.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Non-invasive fibrosis scores progression over time | 5 years
  Change in non-invasive fibrosis scores over time
Incidence of cirrhosis | 5 years
  Incidence of cirrhosis
Incidence of liver-related complications | 5 years
  Incidence of liver-related complications, defined as any of the following: ascites, encephalopathy, gastroesophageal varices, bleeding gastroesophageal varices or hepatocellular carcinoma, whichever occurs first

SECONDARY OUTCOMES:
Fibrosis progression over time | 5 years
  Change in fibrosis score according to liver biopsies over time

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Younossi ZM. Non-alcoholic fatty liver disease - A global public health perspective. J Hepatol. 2019 Mar;70(3):531-544. doi: 10.1016/j.jhep.2018.10.033. Epub 2018 Nov 9. PMID 30414863
- [Result] Lindenmeyer CC, McCullough AJ. The Natural History of Nonalcoholic Fatty Liver Disease-An Evolving View. Clin Liver Dis. 2018 Feb;22(1):11-21. doi: 10.1016/j.cld.2017.08.003. PMID 29128051
- [Result] Patel PJ, Banh X, Horsfall LU, Hayward KL, Hossain F, Johnson T, Stuart KA, Brown NN, Saad N, Clouston A, Irvine KM, Russell AW, Valery PC, Williams S, Powell EE. Underappreciation of non-alcoholic fatty liver disease by primary care clinicians: limited awareness of surrogate markers of fibrosis. Intern Med J. 2018 Feb;48(2):144-151. doi: 10.1111/imj.13667. PMID 29083080
- [Result] Rinella ME, Lominadze Z, Loomba R, Charlton M, Neuschwander-Tetri BA, Caldwell SH, Kowdley K, Harrison SA. Practice patterns in NAFLD and NASH: real life differs from published guidelines. Therap Adv Gastroenterol. 2016 Jan;9(1):4-12. doi: 10.1177/1756283X15611581. PMID 26770262